CLINICAL TRIAL: NCT02906644
Title: Combination Nicotine Patch / Lorcaserin for Smoking Cessation
Acronym: LorNic
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00074741; P50DA027840-06 (NIH)
Record Dates: First submitted 2016-09-15; First posted 2016-09-20 (Estimated); Results first posted 2019-05-07 (Actual); Last update posted 2019-05-07 (Actual); Status verified 2019-05

CONDITIONS: Nicotine Dependence
Keywords: Nicotine addiction; Cigarette smoking; Smoking cessation; lorcaserin; Belviq; Nicotine patches
MeSH Terms: conditions — Tobacco Use Disorder; Cigarette Smoking; Smoking Cessation | interventions — lorcaserin; Tobacco Use Cessation Devices; Nicotine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lorcaserin + Patch (Experimental): Participants will receive lorcaserin (10mg twice a day) and nicotine patches (21mg/24hr) for 14 weeks, at which point the nicotine patch dosage will be reduced to 14mg/24hr for 1 week, followed by 7mg/24hr for 1 week.
  Interventions: Drug: lorcaserin; Drug: nicotine patch
- Patch (Experimental): Participants will receive nicotine patches (21mg/24hr) and placebo lorcaserin for 2 weeks; after 2 weeks participants will begin to receive active lorcaserin (10mg twice a day) along with the nicotine patches for 12 weeks, at which point the nicotine patch dosage will be reduced to 14mg/24hr for 1 week, followed by 7mg/24hr for 1 week.
  Interventions: Drug: lorcaserin; Drug: nicotine patch; Drug: placebo lorcaserin

INTERVENTIONS:
Drug: lorcaserin
  Other Names: Belviq
Drug: nicotine patch
  Other Names: Nicoderm
Drug: placebo lorcaserin
  Other Names: placebo Belviq
  Arms: Patch

SUMMARY:
This study plans to compare the efficacy of the nicotine patch / lorcaserin combination treatment vs. the nicotine patch alone in terms of leading to a reduction in smoking behavior and withdrawal symptoms.

DETAILED DESCRIPTION:
This study proposes to investigate the potential efficacy of a combination of two FDA-approved agents, nicotine patch and lorcaserin, for smoking cessation treatment. The nicotine patch which provides a sustained low dose of nicotine is a nicotine receptor agonist. Lorcaserin, a serotonin 5-hydroxytryptamine receptor 2C (5-HT2C) agonist, is a drug that is FDA-approved for weight loss, and has also recently been shown to be efficacious for smoking cessation. Given that these drugs act through distinct mechanisms it is hoped that the combination will prove more efficacious than either drug alone. It is also hypothesized that the combination will reduce weight gain commonly seen after smoking cessation.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old;
* Smoke an average of at least 10 cigarettes per day;
* Have smoked at least one cumulative year;
* Have an expired air CO reading of at least 10ppm;
* Body weight of >50 kg (110 lbs.)
* Able to read and understand English;
* Express a desire to quit smoking in the next thirty days.

Exclusion Criteria:

* Hypertension (systolic >140 mm Hg, diastolic >100 mm Hg, coupled with a history of hypertension); subjects with no previous diagnosis of hypertension may have a screening blood pressure up to 160/100.
* Hypotension with symptoms (systolic <90 mm Hg, diastolic <60 mm Hg).
* Participants with a history of hypertension may, however, be allowed to participate in the study if the study physician or physician assistant determines that the condition is stable, controlled by medication, and in no way jeopardizes the individual's safety.
* Coronary heart disease, diagnosed by coronary angiogram;
* Lifetime history of heart attack;
* Cardiac rhythm disorder (irregular heart rhythm);
* Chest pain in the last month (unless history, exam, and ECG clearly indicate a non-cardiac source);
* Symptomatic cardiac (heart) disorder (including but not limited to valvular heart disease, heart murmur, heart failure);
* Diagnosis of liver disease or kidney disorder (except kidney stones, gallstones);
* Gastrointestinal problems (e.g. Celiac disease, Crohn's dx Ulcerative Colitis) or disease other than gastroesophageal reflux or heartburn;
* Active ulcers in the past 30 days;
* Currently symptomatic lung disorder/disease (including but not limited to chronic obstructive pulmonary disease (COPD), emphysema, and asthma);
* Brain abnormality (including but not limited to stroke, brain tumor, and seizure disorder);
* Migraine headaches that occur more frequently than once per week;
* Recent, unexplained fainting spells;
* Problems giving blood samples;
* Diabetes (unless controlled by diet and exercise alone and screening glucose is less than 180mg/dcl and HbA1c is less than 7%);
* Current cancer or treatment for cancer in the past six months (except basal or squamous cell skin cancer);
* HIV, Hepatitis B, or Hepatitis C
* History of tuberculosis or recent positive purified protein derivative (PPD) test
* Other major medical condition;
* Current psychiatric disease (with the exception of anxiety disorders, obsessive compulsive disorder (OCD) and ADHD);
* Suicidal ideating (thinking about ways to commit suicide) (within the past 10 years) or lifetime occurrence of attempted suicide;
* Current depression - The Patient Health Questionnaire (PHQ-9) for Depression will be used to screen for current (within 2 weeks) depression. Potential subjects who score >9 (or who score >0 on item #9 ("Thoughts that you would be better off dead, or of hurting yourself in some way") will be excluded from study participation, and, at the discretion of the study physician, referred to appropriate psychiatric treatment;
* Bulimia or anorexia;
* BMI of < 18.5 kg/m2;
* Prior use of fenfluramine or dexfenfluramine
* Use (within the past 30 days) of:

  * Illegal drugs (or if the urine drug screen is positive for tetrahydrocannabinol (THC), Cocaine, Amphetamine, Opiates, Methamphetamines, phencyclidine (PCP), Benzodiazepines, or Barbiturates), Unless recent use of prescription Opiates, Benzodiazepines for management of acute symptoms.
  * Experimental (investigational) drugs;
  * Psychiatric medications including antidepressants (selective serotonin reuptake inhibitors (SSRIs), serotonin and norepinephrine reuptake inhibitors (SNRIs), tricyclic antidepressants (TCAs), monoamine oxidase inhibitors (MAOIs), St. John's Wort), lithium, anti-psychotics or any other medications that are known to affect smoking cessation (e.g. clonidine);
  * Phentermine, triptans, tryptophan, linezolid, dextromethorphan, opiates, tramadol, or dopamine agonists;
  * Any agents that have documented correlation with increased incidence of valvulopathy and/or pulmonary hypertension (e.g., cyproheptadine, trazodone, nefazodone, amoxapine, tricyclic antidepressants, mirtazapine, pergolide, ergotamine, methysergide) (or anticipated use during the study);
  * Smokeless tobacco (chewing tobacco, snuff), pipes or e-cigarettes;
  * Wellbutrin, bupropion, Zyban, Chantix, varenicline, nicotine patch, nicotine replacement therapy or any other smoking cessation aid.
* Concurrent use of a serotonergic agent/combination associated with severe serotonin syndrome (within the past 30 days);
* Use of cigar, cigarillos, pipe, Hookah, dissolvable nicotine, snuff, chewing tobacco more than once per month.
* Use of e-cigarettes once per month or more.
* Self-report of consuming 4 or more alcoholic drinks on 1 or more days per week;
* Significant adverse reaction to lorcaserin or nicotine patch in the past.
* Current participation or recent participation (in the past 30 days) in another smoking study at the investigators Center or another research facility.
* Current participation in another research study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2016-11-08 (Actual); Primary Completion 2018-03-27 (Actual); Study Completion 2018-10-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jed E. Rose, Ph.D., Principal Investigator — Duke University
Locations (1):
- Duke Center for Smoking Cessation, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hartmann-Boyce J, Theodoulou A, Farley A, Hajek P, Lycett D, Jones LL, Kudlek L, Heath L, Hajizadeh A, Schenkels M, Aveyard P. Interventions for preventing weight gain after smoking cessation. Cochrane Database Syst Rev. 2021 Oct 6;10(10):CD006219. doi: 10.1002/14651858.CD006219.pub4. PMID 34611902
- [Derived] Rose JE, Davis JM. Combination Lorcaserin and Nicotine Patch for Smoking Cessation Without Weight Gain. Nicotine Tob Res. 2020 Aug 24;22(9):1627-1631. doi: 10.1093/ntr/ntz149. PMID 31589323

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began on 11/8/2016 and ended on 2/20/2018. Of the 97 subjects (subjs.) consented during this period, 61 subjects met all study criteria, attended the first study visit, were randomized and received study intervention.
Pre-assignment Details: Of the 97 subjs. enrolled, 36 were withdrawn by study staff or withdrew voluntarily from further participation prior to the 1st study visit (V1): 14 did not meet inclusion criteria, 16 met exclusion criteria, 3 were unable to meet study requirements, 2 were excluded due to laboratory values, and 1 was excluded by the medical staff.
Groups:
- Lorcaserin + Patch: Participants will receive lorcaserin (10mg twice a day) and nicotine patches (21mg/24hr) for 14 weeks, at which point the nicotine patch dosage will be reduced to 14mg/24hr for 1 week, followed by 7mg/24hr for 1 week.
  lorcaserin
  nicotine patch
- Patch: Participants will receive nicotine patches (21mg/24hr) and placebo lorcaserin for 2 weeks; after 2 weeks participants will begin to receive active lorcaserin (10mg twice a day) along with the nicotine patches for 12 weeks, at which point the nicotine patch dosage will be reduced to 14mg/24hr for 1 week, followed by 7mg/24hr for 1 week.
  lorcaserin
  nicotine patch
  placebo lorcaserin
Period: First 2 Weeks
Arm/Group | Lorcaserin + Patch | Patch
Started | 31 | 30
Completed | 30 | 27
Not Completed | 1 | 3
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Physician Decision | 1 | 1
Period: Weeks 3 to 14
Arm/Group | Lorcaserin + Patch | Patch
Started | 30 (All participants receiving active Lorcaserin plus nicotine patches starting at the 2nd study visit.) | 27 (All participants receiving active Lorcaserin plus nicotine patches starting at the 2nd study visit.)
Final Study Visit | 17 (All participants receiving only 1 week of 14mg & 1 week of 7mg nicotine patches at this visit.) | 20 (All participants receiving only 1 week of 14mg & 1 week of 7mg nicotine patches at this visit.)
Follow-up (6 Months Post Quit Day) | 14 | 16
Completed | 14 | 16
Not Completed | 16 | 11
Not completed — Withdrawal by Subject | 13 | 7
Not completed — Lost to Follow-up | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lorcaserin + Patch | Patch | Total
Number analyzed (Participants) | 31 | 30 | 61
Age, Continuous [Mean (Full Range); unit: years] | 47 [27 to 65] | 50 [26 to 68] | 49 [26 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 22 | 46
  Male | 7 | 8 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 12 | 8 | 20
  White | 19 | 21 | 40
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 31 | 30 | 61

OUTCOME MEASURES:

1. Primary Outcome: Time-to-lapse
Description: Two weeks after treatment is initiated, with nicotine patch + lorcaserin or nicotine patch alone, but still two weeks prior to the quit day, subjects will be evaluated in a modified version of the McKee Smoking Lapse Task. In this task smokers, who have been abstinent for 2 hours will be provided with the option to smoke at any time, but paid by the minute for remaining abstinent with progressively decreasing payments over an hour.
Time Frame: Week 2 pre quit day
Population: Four participants dropped out of the study and 3 more reported having already quit smoking before the Smoking Lapse Task occurred; therefore, we have lapse data for only 54 participants rather than 61.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Lorcaserin + Patch | Patch
Number analyzed (Participants) | 29 | 25
Minutes | 51.97 (18.331) | 56.44 (12.490)

2. Primary Outcome: Smoking Withdrawal
Description: At the study visit above (two week post treatment initiation but 2 weeks prior to quit day), withdrawal symptoms will be assessed after 2 hours of smoking abstinence using the Shiffman-Jarvik (short form) questionnaire, which consists of 9 items rated from 1 to 7, where 1= not at all, 2= very little, 3= a little, 4= moderately, 5= a lot, 6= quite a lot, and 7= extremely. The 9 items are grouped into 8 subscales: Craving, Negative Affect, Appetite, and Arousal. The range of scores for each subscale will be 1-7, with higher scores indicating more of the withdrawal symptom having been experienced.
Time Frame: Week 2 pre quit day
Population: Four participants dropped out of the study, 3 more reported having already quit smoking before the Smoking Lapse Task occurred, and 1 did not complete the withdrawal questionnaire; therefore, we have lapse data for only 53 participants rather than 61.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lorcaserin + Patch | Patch
Number analyzed (Participants) | 28 | 25
score on a scale
  Craving | 2.81 (1.271) | 2.91 (1.219)
  Negative Affect | 2.15 (0.788) | 2.21 (0.937)
  Arousal | 4.73 (1.014) | 4.72 (1.251)
  Appetite | 3.11 (1.685) | 2.80 (1.607)

3. Secondary Outcome: Number of Participants Reporting Smoking Abstinence
Description: Number of participants who reported continuous four-week abstinence from smoking (weeks 7-10 post target quit date), confirmed by expired air carbon monoxide (CO).
Time Frame: Weeks 7-10 post quit day
Measure: Count of Participants; unit: Participants
Arm/Group | Lorcaserin + Patch | Patch
Number analyzed (Participants) | 31 | 30
Participants | 9 | 10

4. Secondary Outcome: Number of Participants Reporting Tolerability Issues With Lorcaserin + Nicotine Patch Treatment
Description: Tolerability of the lorcaserin + nicotine patch treatment will be assessed by tabulating the number of participants rating side effects > "moderate".
Time Frame: Two Weeks pre and 10 weeks post quit day
Population: Two weeks pre-quit day, all study subjects were switched to taking active lorcaserin for the duration of the study. Twelve participants dropped out of the study prior to the next study visit, therefore side effects data from 2 weeks pre-quit to the end of the study are only available for 49 participants.
Measure: Count of Participants; unit: Participants
Groups:
- Lorcaserin + Nicotine Patch: All participants received active lorcaserin plus nicotine patches starting at Study Visit 2 (two weeks from baseline and two weeks prior to their quit day) after 2 weeks of receiving either active or placebo lorcaserin along with the nicotine patches.
Arm/Group | Lorcaserin + Nicotine Patch
Number analyzed (Participants) | 49
Participants | 26

5. Secondary Outcome: Weight Gain Following Continuous Four-week Abstinence From Smoking
Description: Among smoking-abstinent participants, weight gain relative to baseline will be assessed.
Time Frame: Week 10 post quit day
Population: Two weeks pre-quit day, all study subjects were switched to taking active lorcaserin for the duration of the study. Nineteen participants reported continuous four-week abstinence from smoking (weeks 7-10 post target quit date), confirmed by expired air carbon monoxide (CO).
Measure: Mean (Standard Deviation); unit: weight gain (in lbs)
Arm/Group | Lorcaserin + Nicotine Patch
Number analyzed (Participants) | 19
weight gain (in lbs) | -0.35 (7.203)

6. Secondary Outcome: Number of Participants Reporting 6-month Smoking Abstinence
Description: Number of participants who reported not smoking for the previous seven days when called for 6-month follow-up, confirmed by expired air carbon monoxide (CO).
Time Frame: 6 months post Quit Day
Population: Two weeks pre-quit day, all study subjects were switched to taking active lorcaserin for the duration of the study. Nine participants reported continuous 7-day abstinence from smoking 6 months post quit-day, confirmed by expired air carbon monoxide (CO).
Measure: Count of Participants; unit: Participants
Arm/Group | Lorcaserin + Nicotine Patch
Number analyzed (Participants) | 61
Participants | 9

7. Secondary Outcome: Percentage of Change in Ad Libitum Smoking at End of Week 2
Description: To evaluate the effects of lorcaserin on ad libitum (ad lib) smoking, the percent change in reported number of cigarettes smoked from baseline to the end of week 2 (the day prior to the 2nd study visit) will be calculated.
Time Frame: Week 2 pre quit day
Population: There are insufficient data for 9 participants in the Lorcaserin + Patch group and for 8 participants in the Patch only group (due to participant dropout or incomplete or unreturned diaries) so this analysis excluded those individuals.
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Lorcaserin + Patch | Patch
Number analyzed (Participants) | 22 | 22
percentage of change | -35.58 (0.396) | -47.13 (0.482)

8. Secondary Outcome: Adherence to Lorcaserin + Nicotine Patch Treatment as Indicator of Tolerability
Description: Tolerability of the lorcaserin + nicotine patch treatment will be assessed by calculating adherence scores based on the percentage of days on which the study drugs were taken between visits as reported by participants on diaries.
Time Frame: Two Weeks pre and 10 weeks post quit day
Population: Two weeks pre-quit day, all study subjects were switched to taking active lorcaserin for the duration of the study. Fourteen subjects either dropped out prior to Visit 3 (the first visit after all subjects were on combined treatment) or had missing or incomplete diaries, so data are only available for 47 subjects during this phase of the study.
Measure: Mean (Standard Deviation); unit: percentage of days using study drugs
Arm/Group | Lorcaserin + Nicotine Patch
Number analyzed (Participants) | 47
percentage of days using study drugs | 72.15 (0.339)

ADVERSE EVENTS:
Time Frame: Subjects (subjs.) received (rcvd.) study drugs for 16 weeks. At each study session during this period subjs. completed a questionnaire (quest) about side effects (SE). Subjs. were also told to contact study staff between study sessions if SE were bothersome.
Description: Serious Adverse Events (AE) and other AEs were evaluated for all subjs. who rcvd. nicotine patches and lorcaserin (31) or nicotine patches and placebo (30) at Visit (V) 1, & for all subjs. receiving nicotine patches and lorcaserin at V2 and subsequent visits (56) who completed side effects (SE) quest. Systematic evaluation of SE began at V2 after 2 weeks of study drug use (30 subjs. who had rcvd. nicotine patches and lorcaserin and 27 who had rcvd. nicotine patches and placebo).
Groups:
- Lorcaserin + Patch: Participants will receive lorcaserin (10mg twice a day) and nicotine patches (21mg/24hr) for 14 weeks, at which point the nicotine patch dosage will be reduced to 14mg/24hr for 1 week, followed by 7mg/24hr for 1 week. Group 1 will receive this combined treatment throughout the study; Group 2 will receive the combined treatment after the first 2 weeks of receiving the nicotine patch only (with placebo lorcaserin).
  lorcaserin
  nicotine patch
- Patch (1st 2 Weeks): Participants will receive nicotine patches (21mg/24hr) and placebo lorcaserin for 2 weeks; after 2 weeks participants will begin to receive active lorcaserin (10mg twice a day) along with the nicotine patches for 12 weeks, at which point the nicotine patch dosage will be reduced to 14mg/24hr for 1 week, followed by 7mg/24hr for 1 week.
  lorcaserin
  nicotine patch
  placebo lorcaserin
Arm/Group | Lorcaserin + Patch | Patch (1st 2 Weeks)
All-Cause Mortality (participants affected / at risk) | 0/56 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/56 | 1/27
Other Adverse Events (participants affected / at risk) | 35/56 | 12/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lorcaserin + Patch (N=56) | Patch (1st 2 Weeks) (N=27)
Somnambulism (General disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lorcaserin + Patch (N=56) | Patch (1st 2 Weeks) (N=27)
Fatigue (General disorders) | 12 (14) | 2 (2)
Dizziness/Lightheadedness (General disorders) | 3 (3) | 0 (0)
Insomnia (General disorders) | 4 (5) | 1 (1)
Vivid Dreams (General disorders) | 20 (27) | 9 (9)
Dry Mouth (General disorders) | 7 (13) | 0 (0)
Coughing (General disorders) | 5 (8) | 2 (2)
Nausea (Gastrointestinal disorders) | 3 (3) | 0 (0)
Constipation (Gastrointestinal disorders) | 5 (9) | 0 (0)
Itching at Patch Site (Skin and subcutaneous tissue disorders) | 13 (25) | 4 (4)
Rash at Patch Site (Skin and subcutaneous tissue disorders) | 5 (11) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-12): https://cdn.clinicaltrials.gov/large-docs/44/NCT02906644/Prot_SAP_000.pdf